CLINICAL TRIAL: NCT00649909
Title: Effect of Glucose Control on the Response to Aspirin in Type 2 Diabetic Patients
Status: Completed | Type: Observational
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Principal Investigator, David Varon, Director of coagulation unit, Hadassah Medical Organization
Other Study IDs: 0020-08-HMO-CTIL
Record Dates: First submitted 2008-03-27; First posted 2008-04-01 (Estimated); Last update posted 2017-08-10 (Actual); Status verified 2017-08

CONDITIONS: Diabetes Mellitus, Type II
Keywords: Diabetes Mellitus; Type II; Aspirin; Resistance
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Type 2 diabetic patients with reduced laboratory response to aspirin.(Aspirin Resistance)and with HbA1c >8%.

SUMMARY:
The efficacy of low dose aspirin appears to be substantially lower in diabetic patients, compared to patients without diabetes.

We will perform an observational study where we follow up patients with uncontrolled type 2 Diabetes Mellitus and low response to aspirin (Aspirin Resistance), during a period of 6 months in the diabetic clinic. Our hypothesis is that glucose control will improve the response to aspirin in those patients.

ELIGIBILITY:
Inclusion Criteria

1. Type 2 DM.
2. Patients that take aspirin.
3. Antecubital forearm veins allowing technically good sampling for platelet studies.
4. Reduced Laboratory response to aspirin.
5. HbA1c > 8 %
6. The physician decides that there is an indication for glucose control.

Exclusion Criteria:

1. Acute ischemic stroke, acute coronary syndrome, (myocardial infarction or unstable angina pectoris), or revascularization by PCI or by-pass surgery within the last 6 months.
2. Acute kidney disease or chronic kidney disease with creatinine clearance <30.
3. Acute liver disease or chronic liver disease with severe liver impairment.
4. Need for treatment with anticoagulants, clopidogrel, NSAID's, or thiazolidinediones.
5. Thrombocytopenia (platelet count <150 x 109/L)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Type 2 diabetic patients that take aspirin, from the diabetology clinic.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2008-11; Primary Completion 2010-11 (Actual); Study Completion 2010-11 (Actual)

PRIMARY OUTCOMES:
The outcome measure is the laboratory Aspirin Resistance. | 3 and 6 months.

SECONDARY OUTCOMES:
To determine the incidence of laboratory aspirin resistance in type 2 DM in stable out-patients in the diabetic clinic, and possibly related factors. | On screening visit.

CONTACTS AND LOCATIONS:
Overall Officials: David Varon, MD, Principal Investigator — Hematology Department, Hadassah Medical Organization, Jerusalem, Israel
Locations (1):
- Hadassah Medical Organization, Jerusalem, Israel